CLINICAL TRIAL: NCT00401089
Title: A Placebo-controlled Cross Study of Panax Ginseng in Augmentation of Antipsychotics in 60 Partially Treatment Responsive Patients With Schizophrenia
Brief Title: Efficacy Study of Panax Ginseng to Boost Antipsychotics Effects in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Queen's University (Other); Northern Ontario School of Medicine (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Simon Chiu, University of Western Ontario London Ontario; Research Scientist, Lawson Health Research Institute London Ontario Canada, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R-02-285
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Tardive Dyskinesia; Insulin Resistance; Obesity
Keywords: negative symptoms schizophrenia; Atypical antipsychotics; Neurocognition impairment; obesity risk factor; Diabetes insulin resistance schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Tardive Dyskinesia; Insulin Resistance; Obesity | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginsana-115 (Experimental): Ginsana-115 (Panax Ginseng formulation obtained from Boehringer Ingelheim Pharmaton Inc. Switzerland )is available in oral dosage form of capsules. Two dosages of Ginsana-115 will be tested: 100 mg once daily oral dosage ( 1 100-mg Ginsana-115 capsule) and 200 mg once daily dosage ( 2 100-mg Ginsana-115 capsule). The total duration of each dosage is 8 weeks.
  Interventions: Drug: Panax Ginseng
- Sugar Pill (Placebo Comparator): Placebo capsules formulated identical to the active drug: Ginsana-115 are to be obtained from Boehringer Ingelheim Pharmaton, Switzerland. Two dosages of Placebo capsules will be administered once daily for 8 weeks : a) Placebo 100 mg capsule: 1 placebo capsule daily; b) Placebo 200 mg capsule: 2 placebo-capsule daily
  Interventions: Drug: Panax Ginseng

INTERVENTIONS:
Drug: Panax Ginseng — The standardized extract of Panax Ginseng was formulated by Boehringer Ingelheim Pharmaton, Switzerland and fulfills the criteria of cGMP. Quality control and safety are monitored regularly by Boehringer Ingelheim Pharmaton.
  Other Names: Ginsana-115

SUMMARY:
The objective of the study is to determine whether Panax Ginseng with multiple interactions with key components of brain signaling pathway, can augment the effects of antipsychotics in Schizophrenia. We are primarily interested to examine the actions of Ginseng combined with antipsychotics in improving the ways patients diagnosed with schizophrenia behave in social environment, store, process and retrieve information.

DETAILED DESCRIPTION:
Schizophrenia is a serious mental disorder affecting individuals in multiple ways: behavior control, emotional and information processing and the functional levels conforming to societal norms. Despite recent advances in medication therapy in treating the target symptoms of schizophrenia , subsets of patients diagnosed with schizophrenia continue to exhibit negative symptoms ( social withdrawal,apathy, lack of drive )and cognitive impairment (memory, attention, judgment and reasoning). Recently, there has been interest to explore the efficacy of avenue of dietary and herbal supplements with known pharmacological actions in treatment and prevention of neuropsychiatric disorders, especially bipolar and schizophrenia.

We hypothesize that Panax Ginseng , with multiple interactions with chemical pathways in the brain described as neurotransmitter systems (Dopamine, GABA and NMDA ) can improve the residual symptoms of schizophrenia when added to the antipsychotics currently used in the treatment of schizophrenia. Furthermore, in view of previous studies of Ginseng in enhancing memory , we hypothesize that the standardized formulation of Ginseng (Ginsana-115 from Boehringer Ingelheim-Pharmaton,Switzerland ) will optimize the antipsychotics in cognition impairment and negative symptoms. In the 18-week RCT cross-over study, schizophrenic subjects will be treated with either Ginsana-115 ( 100 mg or 200 mg by oral route) or placebo in a cross-over design. we plan to recruit 60 subjects diagnosed as schizophrenia from the four sites : London-St. Thomas, Ontario, Canada; Kingston Ontario Canada; Thunderbay, Ontario Canada and Middlesex, United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* age 18-65 years
* DSM-IV diagnosis of Schizophrenia
* SANS score greater than 30

Exclusion Criteria:

* Current (past 12 months) substance use disorder
* Except nicotine dependence
* Major medical disorders : hematological disorder
* Chronic active hepatitis, acute hepatitis, cirrhosis of liver, AIDS
* Pregnancy and breast-feeding
* Neurological disorders including epilepsy
* traumatic brain injury
* HAM-D score greater than 24

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-12; Primary Completion 2006-12 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Neuro-Cognitive Screening Test | wk 0, 8, crossover , wk 2, 8
  The battery of neurocognitive tests is to be administered in a computerized format to the subjects at various time intervals
PANSS Positive Negative Syndrome Scale | -wk 2, wk 0, 2, 5,8 crossover wk 2,5,8
  Changes in PANSS is the co-primary outcome measure
SANS | Change from baseline to week 8, cross-over; week 11-week 18.
  We list SANS as the co-primary outcome measure. We cross-validate the changes in SANS with PANSS

SECONDARY OUTCOMES:
HAM-D Hamilton Depression Rating Scale | -wk2, wk0, 2, 5, 8 crossover wk 2, 5, 8
  We will correlate the changes in HAM-D with PANSS changes
BPRS Brief Psychiatric Rating Scale | -wk 2, wk 0, 2,5,8 crossover wk 2, 5, 8
  This is a measure of the global change if any of the psychiatric symptoms during the 18-week period
QLS Quality of Life Scale | wk 0, 8 crossover wk 8
AIMS Abnormal Involuntary Movement Scale | -wk 2, wk 0, 2, 5, 8 crossover wk 2, 5, 8
  We examined whether subjects experienced any changes in dyskinetic movements
SAS Simpson Angus Scale for Extrapyramidal Symptoms | -wk 2, wk 0, 2,5,8 crossover wk 2,5,8
Blood Chemistry Profile: CBC, kidney function,lipid profile, fasting glucose insulin | -wk 2, wk 8 crossover wk 8
  We examined whether the subjects participated in the study experienced any changes in indices of metabolic-metabolic functions
BMI Body Mass index | Change from baseline to end of 18-week period
  BMI will be measured along with anthropometric measures: % total body water;% total fat, % muscle mass

CONTACTS AND LOCATIONS:
Overall Officials: Simon S Chiu, MD PhD, Principal Investigator — Lawson Health Research Institute London Ontario Canada
Locations (4):
- Canada (3):
  - Queen's University, Kingston, Ontario
  - Regional Mental Health Care London, St. Thomas, Ontario
  - Northern Ontario Medical School, Thunder Bay, Ontario
- Northwick Park Hospital, Harrow, Middlesex, United Kingdom